CLINICAL TRIAL: NCT01567683
Title: A Double-blind, Randomized, Single Centre, Vehicle-controlled Study to Evaluate the Safety and Tolerability of a New Topical Formulation Containing 0,09% Imiquimod (Limtop) in Healthy Subjects
Acronym: Limsafe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: LIMTOP-II
Record Dates: First submitted 2012-03-29; First posted 2012-03-30 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Safety and Tolerability of Limtop and vehicle; of Limtop and vehicle
MeSH Terms: interventions — Imiquimod

ARMS (1):
- Limtop solution (imiquimod), Vehicle solution for topical use (Experimental)
  Interventions: Drug: Imiquimod (topical use)

INTERVENTIONS:
Drug: Imiquimod (topical use)

SUMMARY:
This study is designed to assess the tolerability of test product and vehicle in terms of skin reactions during repeated topical applications on healthy skin under controlled conditions on the basis of the international guidelines for testing of skin irritations (FDA Guidance for Industry (1999)).

ELIGIBILITY:
Inclusion Criteria:

1. The written informed consent form (ICF) signed and dated by the subject prior to any study-related activity
2. Generally healthy male or female subjects aged ≥ 18 years
3. Healthy skin in the treatment areas (inner site of forearms) and test field for positive control on the upper arm
4. Skin type I-III (Fitzpatrick)
5. Willingness to actively participate in the study and to comply with the study procedures as defined in the study protocol
6. High probability of a good compliance and orderly completion of the study
7. Female subjects of childbearing potential must use a highly effective method of contraception
8. Negative urine pregnancy test (in female subjects with childbearing potential)

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Known or suspected skin diseases (e.g. acne vulgaris, atopic dermatitis, psoriasis, etc.), which might interfere with the evaluation of the skin reaction at the treatment area or the SLS test field
3. Clinical history suggestive of intolerance, allergies or idiosyncrasies to one of the IMPs or to the ingredients of the products (butyl lactate, isopropyl myristate, propylene glycol, butylated hydroxy anisole) and suspected cross allergies
4. Known skin allergies
5. Known infectious diseases (e.g. HIV, hepatitis) at the discretion of the investigator
6. Insulin dependent diabetes
7. Psychiatric conditions that might limit the participation in the trial and / or that lead to the assumption that the ability to completely understand the consequences of consent is missing
8. Any suspicion of drug and / or alcohol abuse within the past 5 years
9. Any illness or circumstance that could affect the trial purpose in the opinion of the investigator
10. Within 1 week prior to Day 1 and during the whole study any systemic use of antihistamines
11. Within 4 weeks prior to Day 1 and during the entire study no change in any medication with common medical influence on skin perfusion (e.g. beta-blockers)
12. Within 4 weeks prior to Day 1 and during the entire trial any use of systemic medication likely to interfere with the trial purposes (e.g. immune-modulating therapy, corticosteroids, cytotoxics or immunosuppressants)
13. Within 2 weeks prior to Day 1 and during the entire trial: any dermatological medication (drug or medical device) on treatment areas or SLS test field (exceptions: symptomatic treatment of discontinued areas with topical treatments as decided by the investigator)
14. Use of cosmetic product (e.g. creams, moisturizers) in the treatment areas (i.e. inner forearms) or the SLS test field within 5 days prior to Day 1 and throughout the treatment phase (Day 1 to Day 22)
15. Intensive UV-light exposure (e.g. solarium visits) within 4 weeks before Day 1 as well as during the study
16. Moles, tattoos, pigmentation or scars in the application areas (arms) that would influence the visual scoring
17. Participation in another clinical trial within 30 days directly preceding the study, during the entire study, and earlier participation in this study
18. Employees of the study site or of the Sponsor's company

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Proinnovera GmbH Phase I Unit, Münster, Germany